CLINICAL TRIAL: NCT03113825
Title: An Open-Label, Single-Arm, Phase 2 Study of AVB-620 in Women With Primary, Nonrecurrent Breast Cancer Undergoing Surgery
Brief Title: Study of AVB-620 in Women With Primary, Nonrecurrent Breast Cancer Undergoing Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Avelas Biosciences, Inc. (Industry)
Collaborators: RRD International, Inc. (Unknown); Clinipace Worldwide (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVB620-C-002
Record Dates: First submitted 2017-04-04; First posted 2017-04-14 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Primary Invasive Malignant Neoplasm of Female Breast; Carcinoma Breast; Breast Cancer Female; Carcinoma, Ductal, Breast; Stage II Breast Cancer; Stage I Breast Cancer; Stage III Breast Cancer
Keywords: breast carcinoma; DCIS
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Ductal, Breast; Carcinoma, Intraductal, Noninfiltrating | interventions — Drugs, Investigational

STUDY DESIGN:
Intervention Model Description: Period 1 will enroll approximately 35 patients to evaluate conditions to achieve maximal differences in fluorescent signals between malignant and nonmalignant tissue. Period 2 will enroll approximately 120 patients to test dosing and imaging conditions determined in Period 1 and accuracy of AVB-620 imaging data to distinguish between malignant and nonmalignant tissues.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- AVB-620 & Investigational Imaging Device (Experimental): Eligible subjects will receive a single dose of AVB-620 as intravenous infusion before the surgical procedure. During the surgical procedure, fluorescent imaging will be undertaken to distinguish between malignant and nonmalignant tissues.
  Interventions: Device: Investigational Imaging device; Drug: AVB-620

INTERVENTIONS:
Device: Investigational Imaging device — Fluorescence imaging of the of the primary tumor specimen, any secondary breast specimens, and lymph nodes will be performed.
  Other Names: Fluorescent Imaging Camera
Drug: AVB-620 — AVB-620 will be administered IV before the surgical procedure.
  Other Names: Investigational Drug

SUMMARY:
Phase 2, open-label study of AVB-620 in women with primary, nonrecurrent and nonmetastatic breast cancer undergoing surgery.

DETAILED DESCRIPTION:
Phase 2, open-label study of AVB-620 in women with primary, nonrecurrent, nonmetastatic breast cancer undergoing either a lumpectomy with simultaneous sentinel lymph node biopsy (SLNB) or axillary lymph node dissection (ALND), or a mastectomy and simultaneous ALND. AVB-620 is a synthetic protease-activated peptide dye conjugate administered intravenously for the fluorescence detection and localization of potentially malignant tissue in primary tumor, tumor margins, or lymph nodes. A fluorescence image will be displayed on a monitor and will assist the surgeon to assess potentially cancerous tissue within the primary tumor site, tumor margins, or in lymph nodes which drain the primary tumor site.

Eligible patients will receive a single dose of AVB-620 by IV infusion up to 24 hours prior to breast surgery.

The study will evaluate the effect of timing of AVB-620 administration relative to surgery on the fluorescence and the accuracy of the AVB-620 imaging data to distinguish between malignant and nonmalignant tissues.

ELIGIBILITY:
Inclusion Criteria:

* DCIS or Stage I-III primary invasive carcinoma of the breast
* Primary surgical treatment is lumpectomy + SLNB or ALND --or-- mastectomy + ALND
* Signed written informed consent
* At least 18 years of age
* ECOG performance status 0 to 2
* Life expectancy of at least 6 months
* Total bilirubin ≤ 2 mg/dL
* AST/SGOT and ALT/SGPT ≤ 2.5 X ULN
* Negative serum pregnancy test and using medically acceptable form of contraception if of child bearing potential
* LVEF within normal limits if patient received prior anthracycline therapy [Period 1].

Exclusion Criteria:

* Recurrent ipsilateral breast cancer
* Prior neoadjuvant chemotherapy, endocrine therapy, or biologic therapy for current breast cancer [Period 2]
* Prior neoadjuvant chemo or biologic therapy for current breast cancer within 4 weeks prior to planned surgery [Period 1]
* Open surgery in ipsilateral breast within 1 year.
* Prior malignancy, other than breast cancer, active within the last 6 months
* Prior radiation therapy to the chest [Period 2]
* Radiation therapy to ipsilateral breast [Period 1]
* Abnormal cardiac rhythm not controlled with medication; Hx of stroke within 1 year; Hx of coronary events and/or heart failure within 1 year.
* Diagnosis of autoimmune disorder, including RA, SLE, or Sjogren's syndrome
* Hx of drug-related anaphylactic reactions, severe allergic reactions related to drug; active diagnosis of uncontrolled airway hyperactivity, uncontrolled asthma, or asthma requiring oral corticosteroids.
* Hx of drug-induced acute tubular necrosis.
* Chronic renal failure or current evidence of moderate to severe renal impairment.
* Current diagnosis of any other active or clinically significant nonbreast cancer
* Received systemic investigational drug within 6 weeks prior to AVB-620 administration or has received AVB-620 previously.
* Pregnant or breast feeding or plans to become pregnant within 6 months of AVB-620 administration.
* Unresolved acute toxicity from prior anticancer therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with DCIS or Stage I-III breast cancer who are undergoing lumpectomies or mastectomies and sentinel lymph node biopsies or axillary lymph node dissection.
Enrollment: 92 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2020-04-08 (Actual); Study Completion 2020-11-18 (Actual)

PRIMARY OUTCOMES:
Determine the accuracy of AVB-620 imaging data to distinguish between malignant and nonmalignant tissues. | 1 month
  Determine the accuracy of AVB-620 in correlating image-identified malignant breast or lymph node tissue with pathology findings in breast cancer patients.

SECONDARY OUTCOMES:
Safety of AVB-620 as assessed by incidence of adverse events and abnormal laboratory values. | 1 month
  Evaluate the safety and tolerability of a single AVB-620 infusion in women undergoing breast cancer surgery.
Identify malignant tissue types that provide the most robust fluorescence response compared to non-malignant tissue. | 1 month
  Measure fluorescence intensity differences between malignant and non-malignant tissue to identify best responding tissue type.
Evaluate timing of AVB-620 administration on optical fluorescence characteristics | 1 month
  Further evaluate the effect of the timing of AVB-620 administration on the optical fluorescence characteristics

OTHER OUTCOMES:
Evaluate imaging techniques and conditions | 1 month
  Evaluate the impact of changes in intraoperative imaging techniques and conditions in distinguishing malignant from nonmalignant tissue compared to pathological assessment.
Evaluate methods for image analysis and display | 1 month
  Evaluate and refine methods and criteria by which images are analyzed and displayed
Evaluate breast cancer patient suitability for AVB-620 imaging | 1 month
  Evaluate which breast cancer patients are most suitable for AVB-620 imaging
Determine re-excision rates | 4 weeks
  Determine the planned and actual re-excision rates within 4 weeks after AVB-620 administration.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Chen, MD, MBA, Study Director — Avelas Biosciences, Inc.
Locations (13):
- United States (13):
  - UCSD, San Diego, California
  - Medstar Washington Hospital, Washington D.C., District of Columbia
  - Mayo Clinic Jacksonville -- Center for Breast Health, Jacksonville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Advocate Good Shepherd Hospital, Barrington, Illinois
  - William Beaumont Hospital, Royal Oak, Michigan
  - UNLV School of Medicine, Las Vegas, Nevada
  - Roswell Park Cancer Institute, Buffalo, New York
  - Montefiore Einstein Center for Cancer Care, The Bronx, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Ohio State University, James Cancer Center, Columbus, Ohio
  - Roper St. Francis Hospital, Charleston, South Carolina
  - Swedish Cancer Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No